CLINICAL TRIAL: NCT07257224
Title: Post-market Clinical Follow-up Study of an Isotonic Saline Solution to Manage Nasal Congestion in Case of Flu Symptoms, Colds, Allergic Rhinitis and Rhinosinusitis in Infants and Toddlers
Acronym: Nasal Baby
Status: Not yet recruiting | Type: Observational
Sponsor: Laboratoires Quinton International S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: NASBA01
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Nasal Congestion; Common Cold; Allergic Rhinitis; Rhinosinusitis; Flu Symptom
Keywords: infants; toddlers; Upper Respiratory Tract Infections; Pediatric nasal spray; nasal spray; Seawater isotonic solution; Post-market clinical follow-up (PMCF)
MeSH Terms: conditions — Nasal Obstruction; Common Cold; Rhinitis, Allergic; Rhinosinusitis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Nasal Congestion Cohort: Infants and toddlers (3 to 48 months) with nasal congestion due to flu, colds, allergic rhinitis, or rhinosinusitis. All participants will use the CE-marked nasal spray according to its Instructions for Use.
  Interventions: Device: Quinton Medical Nasal Health Baby®

INTERVENTIONS:
Device: Quinton Medical Nasal Health Baby® — CE-marked Class IIa isotonic seawater nasal spray intended for nasal hygiene and relief of nasal congestion in infants and toddlers. In this study, the device will be administered according to its Instructions for Use, up to 6 applications per day, for a maximum of 14 days. Participants will be evaluated at Day 2, Day 5, and Day 14 for symptom relief, nasal discharge clearance, breathing improvement, sleep quality, and safety outcomes.

SUMMARY:
The goal of this observational post-market clinical follow-up study is to evaluate the safety and performance of the CE-marked nasal spray in the management of nasal congestion in case of flu, colds, allergic rhinitis and rhinosinusitis in infants and toddlers aged 3 to 48 months at day 5 post-enrolment. Enrolment does not require establishing a medical diagnosis; eligibility is based on guardian-reported nasal congestion consistent with lay use of the device.

Participants will be:

* Evaluated by a healthcare professional for eligibility.
* Receive treatment with the CE-marked nasal spray according to its Instructions for Use, for up to 14 days.
* Have their legal guardians report symptom severity and improvement using standardized scales (Visual Analog Scale) during follow-up visits on Day 2, Day 5, and Day 14 and device usability on Day 14.

This study does not include a comparison group and reflects real-world use of the device in routine pediatric care.

DETAILED DESCRIPTION:
This is a prospective, observational, post-market clinical follow-up (PMCF) study designed to collect real-world data on the safety and performance of an isotonic seawater nasal spray in the management of nasal congestion in case of flu, colds, allergic rhinitis and rhinosinusitis in infants and toddlers aged 3 to 48 months.

The device is CE-marked as a Class IIa medical device under MDR 2017/745 and is already commercially available. Therefore, no investigational assignment or randomization is required. Participants will use the marketed device according to its Instructions for Use.

The study will enroll children who meet defined inclusion and exclusion criteria and whose legal guardians provide informed consent. Follow-up assessments are scheduled at Day 2, Day 5, and Day 14, with the primary evaluation point at Day 5. Legal guardians will report outcomes such as nasal congestion relief, secretion clearance, and breathing improvement using validated Visual Analog Scales (VAS). Safety data, including adverse events, will be collected throughout the 14-day period.

The primary objective is to confirm short-term safety and performance at Day 5. Secondary objectives include assessing sustained effects and safety through Day 14, subject legal guardian's satisfaction, and impact on sleep quality.

This study is being conducted at two centers in Spain and is expected to recruit over a 10-month period, with a total study duration of approximately 11 months.

Results will provide additional clinical evidence to support the continued safe and effective use of isotonic seawater nasal sprays in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants / toddlers aged 3 to 48 months (inclusive) at the time of enrolment.
* Subjects with flu, cold, allergic rhinitis or rhinosinusitis as reported by their legal guardian(s) and/or medical history.
* Subjects presenting at least moderately bothersome nasal congestion (blocked or stuffy nose) as reported by their legal guardian(s) and/or medical history and confirmed by the site investigator through non-diagnostic inspection.
* Subjects suitable for nasal hygiene treatment with the study device according to its IFU.
* Subjects with nasal congestion symptoms that began within 48 hours prior to enrolment.
* Subjects whose legal guardian(s) signed written informed consent on their behalf to participate in the study.
* Subject whose legal guardian(s) are willing and able to follow the IFU and comply with all study procedures.

Exclusion Criteria (if any severe symptoms are seen in the subject, the guardian will be advised to seek medical evaluation by the subject's physician):

* Subjects with known hypersensitivity or intolerance to seawater or any of its natural mineral components (e.g., sodium, chloride, magnesium) as reported by their legal guardian(s) and/or medical history.
* Subjects showing severe symptoms such as persistent fever (>38°C), severe cough, ear pain, or respiratory distress, as reported by their legal guardian(s) and/or medical history.
* Subjects whose legal guardian(s) and/or medical history report any ongoing medical diagnosis or treatment for acute infection or chronic respiratory disease (e.g., asthma, pneumonia, laryngotracheobronchitis, sinusitis, etc.).
* Subjects whose legal guardians(s) and/or medical history report any type of immunodeficiency.
* Subjects whose legal guardian(s) and/or medical history report a neurological condition that may affect respiratory functioning.
* Subjects with visible nasal injury, wounds or bleeding, or any condition that may contraindicate the use of the study device according to the device IFU.
* Subjects who are currently participating or have participated in another clinical investigation within the last 30 days prior to enrolment.
* Subjects using saline nasal drops or nasal sprays or pumps other than the study product within 12 hours prior to the time of enrolment or during the study.
* Subjects using the study product within 24 hours prior to the time of enrolment in the study.
* Subject using antibiotics, antivirals, intranasal medications, decongestants, antihistamines, mucolytics, echinacea, combination cold formulas, supplements containing ≥ 10 mg zinc that could influence symptom scores within 12 hours prior to the time of enrolment or during the study.

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and toddlers aged 3 to 48 months, both male and female, presenting with nasal congestion associated with flu, common cold, allergic rhinitis, or rhinosinusitis, recruited from pediatric clinical practices and pediatric physiotherapy clinics.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety - Treatment-related AEs and SAEs at Day 5 Performance - Improvement in nasal congestion improvement indicators at Day 5 | Baseline to Day 5
  Safety: Occurrence of Treatment-related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) at day 5 post-enrolment with daily device use as per the device Instructions for Use (IFU).
  Performance: Relief of nasal congestion, improvement in nasal discharge clearance and improvement of breathing at day 5 post-enrolment with daily device use as per IFU assessed by VAS (0-10) by legal guardian(s).
Functioning - Symptom improvement at Day 5 | Baseline to Day 5
  Change in participant caregiver-reported symptom severity (nasal congestion, nasal discharge clearance, and breathing) using a Visual Analog Scale (VAS, 0-10) from baseline to Day 5 with daily treatment with Quinton Medical Nasal Health Baby® as per its Instructions for Use.

SECONDARY OUTCOMES:
Safety - AEs, TRAEs, and SAEs up to Day 14 | Baseline to Day 14
  Number and proportion of participants experiencing any adverse events (AEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs) during the 14-day study period.
Functioning - Symptom improvement and participant guardian-reported outcomes up to Day 14 | Baseline to Day 14
  Change in participant guardian-reported symptom severity (nasal congestion, secretion clearance, and breathing) at Days 2, and 14 compared to baseline using VAS (0-10); time to onset of perceived symptom relief; frequency of analgesic use; improvement of sleep quality at Days 2, 5 and 14 compared to baseline; and guardian's satisfaction at Day 14 using a 7-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica Uner, Alicante
  - Nombre de Mujer, Alicante

IPD SHARING:
Plan to Share IPD: No
The sponsor does not plan to share individual participant data with other or external researchers. All data will be pseudonymised and assigned a study-specific code before being entered into an electronic data collection system. Each site will have access only to the data of participants recruited at their own centre.